CLINICAL TRIAL: NCT05568030
Title: Evaluation of the Efficacy of a Single Brief Intervention of Mindfulness to Reduce Stress Response in a Social Stress Task Paradigm
Acronym: SBST_FMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Chantal Berna, Professor, University of Lausanne Hospitals
Allocation: Not Applicable | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CER-VD 2022-01316
Record Dates: First submitted 2022-09-01; First posted 2022-10-05 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Mindfulness; Fibromyalgia; Stress
MeSH Terms: conditions — Fibromyalgia | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness (Experimental)
  Interventions: Behavioral: Mindfulness
- Psycho-education (Active Comparator)
  Interventions: Behavioral: Psycho-education

INTERVENTIONS:
Behavioral: Mindfulness — One session of a 20 minute mindfulness recording, based on standardised script, focused on stress management.
  Arms: Mindfulness
Behavioral: Psycho-education — One session of a 20 minute recording, based on standardised script, focused on psychophysiological stress response description.
  Arms: Psycho-education

SUMMARY:
This study is a double-blinded randomized controlled trial with two arms, comparing a recorded mindfulness intervention to a control psycho-education audio. It is a monocentric study that will take place in Centre Hospitalier Universitaire Vaudois (CHUV), a primary teaching hospital in Lausanne, Switzerland.

Patients will be randomized 1:1 to the brief mindfulness intervention vs neutral audio intervention. The investigators involved in recruitment and testing will be blind to the intervention condition. A collaborator that is not involved in this study will prepare a coded randomized sequence of audio assignments, uploaded in Redcap. The audio will be played on a laptop or mp-player with a noise cancelling headset.

ELIGIBILITY:
Inclusion Criteria:

* We plan to recruit adult female patients (>18 years old) suffering from fibromyalgia (FMS), with chronic pain (more than 6 months), willing and able to give informed consent. Specifically, patients must fulfil the criteria of the American College of Rheumatology (2010) by having the following combination of scores at the widespread pain index (WPI) and the severity score (SS) :
* WPI score is ≥7 and the SS score is ≥ 5 OR
* WPI score is comprised between 3 to 6 and the SS score ≥9
* And no other condition explaining the painful syndrome

Exclusion Criteria:

* Insufficient French language skills
* Unstable psychiatric co-morbidity: major depression with current suicidal risk, unstable psychotic disorder, unstable psychotropic medication (stable=more than 3 month under the same dose).
* Somatic co-morbidity that could interfere with physiological monitoring/stress tolerance: such as cardiac malformation, recent myocardial dysfunction, cardiac transplantation, or cardiac treatment (pacemaker, antiarrhythmic drugs, muscarinic receptor blockers, ACE inhibitors or any that would induce a modification in HR)
* Contraindication to sensors positioning (local skin damage or allergies)
* Substance use disorder (alcohol, drugs).
* Refusal to listen to an audio recording of mindfulness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Perceived stress reactivity | Within 3 hours
  The primary outcome is the variation of perceived stress level along the task. A 2-way repeated-measures ANOVA will be conducted to compare the stress reactivity of patients receiving the mindfulness intervention and the control intervention.
  Perceived stress will be measured using visual analog scales from 0 to 10, 0 meaning no stress perceived and 10 meaning the highest stress perceived.

SECONDARY OUTCOMES:
Heart rate variability | Within 3 hours
  Heart rate variability will also be measured using a NeXus-10 MKII, Mindmedia with 3 electrodes.
  A 2-way repeated-measures ANOVA will be conducted to compare the heart rate variability of patients receiving the mindfulness intervention and the control intervention.
Respiration rate | Within 3 hours
  Respiration rate will also be measured using a NeXus-10 MKII, Mindmedia with a thoracic belt.
  A 2-way repeated-measures ANOVA will be conducted to compare the respiration rate of patients receiving the mindfulness intervention and the control intervention.
Oxygen saturation | Within 3 hours
  Oxygen saturation will also be measured using a NeXus-10 MKII, Mindmedia with a pulse oximeter probe.
  A 2-way repeated-measures ANOVA will be conducted to compare the oxygen saturation of patients receiving the mindfulness intervention and the control intervention.
Electrodermal activity | Within 3 hours
  Electrodermal activity will also be measured using a NeXus-10 MKII, Mindmedia with two fingertips electrodes.
  A 2-way repeated-measures ANOVA will be conducted to compare the electrodermal activity of patients receiving the mindfulness intervention and the control intervention.
Cerebral activity | Within 3 hours
  Cerebral activity will also be measured using a 6-electrodes headband electroencephalogram (Dreem headband, Dreem SAS).
Salivary cortisol concentrations | Within 3 hours
  Salivary cortisol concentration will also be collected using a mouth cotton swab. A 2-way repeated-measures ANOVA will be conducted to compare the salivary cortisol concentrations of patients receiving the mindfulness intervention and the control intervention.
Blood catecholamine levels | Within 3 hours
  Blood catecholamine levels will also be collected using a venous line on the non-dominant arm for repeated blood collection. A 2-way repeated-measures ANOVA will be conducted to compare the blood catecholamine levels of patients receiving the mindfulness intervention and the control intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Berna, Prof, Principal Investigator — Centre de médecine intégrative et complémentaire, CHUV
Locations (1):
- Centre de Médecine Intégrative et Complémentaire, CHUV, Lausanne, Canton of Vaud, Switzerland